CLINICAL TRIAL: NCT06071546
Title: Pre-market Monocentric Cross-sectional Clinical Investigation of MAIA on Healthy Subjects and Patients With Retinal Pathology: Agreement With MAIA 2013 EDITION Microperimeter and Repeatability Evaluation
Brief Title: Clinical Investigation of a New Version of MAIA Microperimeter on Healthy Subjects and Patients With Retinal Pathology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centervue SpA (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MAIA_003_MAG
Record Dates: First submitted 2023-09-22; First posted 2023-10-06 (Actual); Last update posted 2024-08-13 (Actual); Status verified 2024-08

CONDITIONS: Healthy Eyes; Retinal Diseases
MeSH Terms: conditions — Retinal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Main arm (Experimental): * one microperimetric examination with MAIA, one microperimetric examination with MAIA 2013 EDITION for agreement evaluation;
  * one additional microperimetric examination with MAIA and one additional microperimetric examination with MAIA 2013 EDITION for repetability evaluation.
  Interventions: Device: MAIA

INTERVENTIONS:
Device: MAIA — MAIA is a visual field testing device combining visual field tests, fixation loss correction by a real-time retinal tracker and confocal TrueColor fundus imaging (P/N AHMACME001)

SUMMARY:
The purpose of this pre-market, monocentric cross-sectional study is to evaluate the clinical usefulness of a new version of the MAIA device (MAIA) through an agreement with the established version of the MAIA microperimeter (MAIA 2013 EDITION). Moreover, the study aims to evaluate MAIA test-retest repeatability in comparison with MAIA 2013 EDITION and to evaluate MAIA safety and adverse events. These purposes will be achieved by collecting data of healthy subjects and patients with retinal pathology. All participants will undergo repeated microperimetric examinations with both devices during one single visit.

ELIGIBILITY:
Healthy Subjects

Inclusion Criteria:

* Age: 18-90 years old;
* BCVA ≥ 0.8 Decimal;
* Equivalent spherical refraction between -12D and +6D; astigmatism within 2D;
* IOP ≤ 21 mmHg;
* Clinically normal appearance of the optic nerve head (examined with Spectralis OCT);
* Clinically normal appearance of the macula (examined with Spectralis OCT);
* No ocular pathologies, trauma, surgeries;
* Absence of pathologies that can affect visual field;
* No use of drugs inferfering with the correct execution of perimetry;

Exclusion Criteria:

* Glaucoma or glaucoma suspect diagnosis;
* IOP ≥ 22 mmHg;
* Presence or history of disc hemorrhage;
* Presence of amblyopia;
* Nystagmus or poor fixation;
* Previous laser or any ocular surgery, including uncomplicated cataract surgery performed within 6 months before enrollment;
* Any active infection of anterior or posterior segments;
* Subjects with significant ocular media opacities;
* Evidence of diabetic retinopathy, diabetic macular edema, or other retinal disease;
* Use of any drug that can interfere with the correct execution of microperimetry or that would produce visual field loss;
* Unable to tolerate ophthalmic imaging;
* Claustrophobia;
* Inability to provide informed consent.

Patients with retinal pathology

Inclusion Criteria:

* Age: 18-90 years old;
* BCVA ≥ 0.1 Decimal;
* Equivalent spherical refraction between -12D and +6D; astigmatism within 2D;
* Diagnosis of any type of retinal disease by investigator based on fundoscopy and Spectralis OCT for which microperimetry is indicated;

Exclusion Criteria:

* Any ocular surgery, with the exception of uncomplicated cataract surgery performed at least 6 months before enrollment;
* Subjects unable to tolerate ophthalmic imaging;
* Nystagmus;
* Subjects with significant ocular media opacities;
* Use of any drug that can interfere with the correct execution of microperimetry or that would produce visual field loss;
* Claustrophobia;
* Inability to provide informed consent;
* Vulnerable subjects according to the investigator's judgement.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 68 (Actual)
Dates: Start 2023-10-17 (Actual); Primary Completion 2024-07-12 (Actual); Study Completion 2024-07-12 (Actual)

PRIMARY OUTCOMES:
To evaluate the limits of agreement between MAIA and MAIA 2013 EDITION for threshold sensitivity values. | 1 day
  Agreement will be quantified by using the method proposed by Bland and Altman [1,2,3], estimating the 95%-Limits of Agreement (LoA) of the difference of threshold sensitivity values.
  The acceptance criteria for agreement between MAIA and MAIA 2013 EDITION is that MAIA's 95% LoA limits are within MAIA 2013 EDITION repeatability limits.
  1. Bland JM, Altman DG (1986) Statistical methods for assessing agreement between two methods of clinical measurement. Lancet 1(8476):307-10.
  2. Bland JM, Altman DG (1999) Measuring agreement in method comparison studies. Statistical Methods in Medical Research 8:135-160
  3. Bland JM, Altman DG (2007), Agreement Between Methods of Measurement with Multiple Observations Per Individual, Journal of Biopharmaceutical Statistics 17:571-82

SECONDARY OUTCOMES:
To assess the repeatability limits of retinal threshold sensitivity values obtained with MAIA | 1 day
  The acceptance criteria is that the 95% LoA limits for MAIA are at least as narrow as MAIA 2013 EDITION repeatability limits.
To assess the avoidance of Serious Adverse Device Effects with MAIA | through study completion (expected duration: 3 months)
  During the clinical investigation, adverse events will be documented, investigated and reported according to the provisions of applicable reporting guidelines, following their criteria and timelines

CONTACTS AND LOCATIONS:
Overall Officials: Maximilian Pfau, PD Dr. med., Principal Investigator — Universitätsspital Basel, Augenklinik
Locations (1):
- Universitätsspital Basel, Augenklinik, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ansari G, Giudici NL, Cancian G, Rossouw P, Rui C, Rosso A, Gazzina S, Feltgen N, Pfau K, Pfau M. Validation and Repeatability of Differential Light Sensitivity Measurements with the Novel MAIA Microperimetry Device. Ophthalmol Sci. 2025 Jul 16;5(6):100886. doi: 10.1016/j.xops.2025.100886. eCollection 2025 Nov-Dec. PMID 40980023